CLINICAL TRIAL: NCT00516009
Title: Efficacy of Intravenous Dexamethasone for Acute Disc Herniation-Induced Sciatica
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-7-247S
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: RADICULAR PAIN
Keywords: RADICULAR PAIN; DISC HERNIATION; DEXAMETHASONE; VAS
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 TREATMENT GROUP (Experimental): 20 PATIENTS WILL RECEIVE DEXAMETHASONE 30 MG IV 3 DAYS AND 20 AND 10 MG FOR THE OTHER TWO DAYS
  Interventions: Drug: DEXAMETHASONE
- 2 (Placebo Comparator): 20 PATIENTS WILL RECEIVE PLACEBO FOR 5 DAYS
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: DEXAMETHASONE
  Arms: 1 TREATMENT GROUP
Other: PLACEBO
  Arms: 2

SUMMARY:
Acute low back pain is one of the most common reasons for all physician visits(1). Phospholipase A2 (PLA2), a potent inflammatory mediator, has demonstrated to be released by discs following injury(4). Clinical practice and animal research suggest that lumbar radicular pain is the result of inflammation of the nerve root in the epidural space(5). The study will evaluate the efficacy of intravenous Dexamethasone for acute disc herniation-induced sciatica. 40 patients aged 18 years or older, who will be transferred to the emergency room due to sciatic pain will be blindly randomized to receive Dexamethasone 30 mg IV for 3 days an tapering off, 10 mg daily, or normal saline. 20 patients will be in each group. The patients will continue their standard care during the study period. Follow up will last for 3 months. Mann-Whitney test will be used for parametric correlation, Wilcoxon for numeral and x² for categorial variables. Dexamethasone IV can help physicians in treating patients with acute sciatic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older presented with acute radicular pain for less than 6 weeks.

Exclusion Criteria:

* Patient with acute infection,
* Psychiatric disorder,
* Uncontroled diabetes,
* Uncontrolede hypertension,
* Severe congestive heart failure,
* Cauda equina syndrome,
* Moderate or severe motor deficit,
* Primary spinal stenosis,
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: RADI SHAHIEN, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Neurology Unit - Ziv Mc, Safed, Israel

REFERENCES:
- [Background] Atul TP and Abna AO. Diagnosis and Management of Acute Low Back Pain. American Family Physician. Published by The American Academy of Family Physicians, March 15, 2000.
- [Background] Engstrom JW. Back and neck pain. In: Kasper DL, Braunwald E, Fauci A, et al, eds. Harrison's Principles of Internal Medicine. 16th ed. New York: McGraw-Hill; 2005: 94-104.
- [Background] Patel N. Surgical disorders of the thoracic and lumbar spine: a guide for neurologists. J Neurol Neurosurg Psychiatry. 2002 Sep;73 Suppl 1(Suppl 1):i42-8. doi: 10.1136/jnnp.73.suppl_1.i42. No abstract available. PMID 12185261
- [Background] Gerard Malanga. Corticosteroid in the Treatment of Acute Low Back Pain. www.spineuniverse.com.
- [Background] Boqing C and Patrick M. Epidural Steroid Injections. August 11, 2005; www.emedicine.com.
- [Background] Finckh A, Zufferey P, Schurch MA, Balague F, Waldburger M, So AK. Short-term efficacy of intravenous pulse glucocorticoids in acute discogenic sciatica. A randomized controlled trial. Spine (Phila Pa 1976). 2006 Feb 15;31(4):377-81. doi: 10.1097/01.brs.0000199917.04145.80. PMID 16481946
- [Background] Korhonen T, Karppinen J, Malmivaara A, Autio R, Niinimaki J, Paimela L, Kyllonen E, Lindgren KA, Tervonen O, Seitsalo S, Hurri H. Efficacy of infliximab for disc herniation-induced sciatica: one-year follow-up. Spine (Phila Pa 1976). 2004 Oct 1;29(19):2115-9. doi: 10.1097/01.brs.0000141179.58778.6c. PMID 15454701
- [Background] Korhonen T, Karppinen J, Paimela L, Malmivaara A, Lindgren KA, Bowman C, Hammond A, Kirkham B, Jarvinen S, Niinimaki J, Veeger N, Haapea M, Torkki M, Tervonen O, Seitsalo S, Hurri H. The treatment of disc-herniation-induced sciatica with infliximab: one-year follow-up results of FIRST II, a randomized controlled trial. Spine (Phila Pa 1976). 2006 Nov 15;31(24):2759-66. doi: 10.1097/01.brs.0000245873.23876.1e. PMID 17108825